CLINICAL TRIAL: NCT04452539
Title: Gender Influence on Mortality and Major Morbidity After Pediatric Cardiac Surgery.
Brief Title: Gender Influence on Morbi-mortality in Pediatric Cardiac Surgery.
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Head, Department of Anesthesiology, Brugmann University Hospital
Other Study IDs: CHUB_GENDERPED
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Pediatric Cardiac Surgery; Gender
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paediatric cardiac surgery patients: All patients undergoing paediatric cardiac surgery
  Interventions: Procedure: Paediatric cardiac surgery

INTERVENTIONS:
Procedure: Paediatric cardiac surgery — All patients undergoing paediatric cardiac surgery

SUMMARY:
Recent studies show an important influence of gender on inflammatory reactions. Cardiac surgery is associated with a major systemic inflammatory response. The investigators want to evaluate the gender influence on morbi-mortality in pediatric cardiac surgery patients.

DETAILED DESCRIPTION:
Gender plays an important role in the inflammatory response. This is due to hormonal influences, but also different genetic regulation of pro-inflammatory cytokines, as nuclear facto kapp B. it is also know that cardiac surgery, especially under cardiopulmonary bypass, is associated with a major inflammatory response. This response is even more marked in pediatric cardiac surgery. The investigators hypothesise that there is a gender influence on mortality and major morbidity in paediatric patients undergoing cardiac surgery. The investigators will do a retrospective cohort study, analysing the local database of all paediatric cardiac surgery cases from jan 2006 to dec 2019. Primary outcome will be any difference in mortality and /or major morbidity according to gender.

Statistical analysis:

The investigators will use a propensity score on 11 pre-operative variables clinically judged relevant. Both group will be matched until a absolute standardised difference < 15% is obtained. This type of matching, contrary to a P value, is independent of sample size. Variables will be presented as mean, standard deviation or percentage for frequency distributions. After propensity score matching, logistic regressions will be performed on binary variables and linear regressions on continuous variables. A Bonferroni correction will be used for multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing paediatric cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* Jehova's witness

Max Age: 16 Years | Sex: All
Age Groups: Child
Study Population: All patients undergoing paediatric cardiac surgery with cardiopulmonary bypas at our institution from jan 2006 to dec 2019.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Mortality | Beginning of the operation until 5 days postop
  Mortality in paediatric cardiac surgery
Morbidity | Beginning of the operation until 5 days postop
  Major morbidity in paediatric cardiac surgery, defined as at least 2 of the following conditions: Respiratory failure (mechanical ventilation > 90h), prolonged inotropic support (> 5 mcg/kg/min of dobutamine for more than 48h postop), renal insufficiency (Drop in glomerular filtration rate > 75% compared to preop values)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Schmartz, MD, Principal Investigator — CHU Brugmann
Locations (1):
- Hôpital Universitaire des Enfants Reine Fabiola, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No